CLINICAL TRIAL: NCT03582605
Title: Antibiotic Prophylaxis Prior to the Insertion of Orthodontic Mini-screw Implants: a Randomized Controlled Trial
Brief Title: Antibiotics Prior to Mini-screw Implant Insertion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Byron Schroeder, DDS, Saint Louis University Orthodontic Resident, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 29379
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Inflammation at Mini-screw Insertion Site; Mobility, Mini-screw
Keywords: antibiotics; prophylaxis; temporary anchorage devices; mini-screw implants; TADs; MSIs; failure rate
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind randomized control trial in which half the participants will be given two grams of amoxicillin in capsule form, prepared by a pharmacist, and the other half will be given a placebo in capsule form, prepared by a pharmacist, 1 hour prior to MSI placement. Sealed envelopes containing either antibiotics or placebo capsules will be given to patients, with only the research committee chair knowing which patients are in the control group (placebo) and which are in the experimental group (antibiotics). Test subjects will be followed for 1 month (T1), 3 months (T2), 6 months (T3) following placement of MSIs.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Amoxicillin and the placebo (glucose) will be prepared in capsule form by a pharmacist and made to look identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): All participants will be weighed. This group will receive a placebo (glucose) 1 hour prior to insertion of mini-screw implants.
  Interventions: Drug: Placebo oral capsule
- Experimental Group (Experimental): All participants will be weighed so that appropriate dosing can be ensured and will receive 2 grams of Amoxicillin 1 hour prior to mini-screw insertion. Patients weighing less than 40 kg will be given 50mg/kg of Amoxicillin.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — see previous descriptions
  Arms: Experimental Group
Drug: Placebo oral capsule — see previous descriptions
  Arms: Control Group

SUMMARY:
The investigators plan to use amoxicillin in capsule form, prepared by a pharmacist, for antibiotic prophylaxis to decrease the failure rate of mini-screw implants temporarily placed in the palate of patients involved in Phase II orthodontics treatments. The mini-screws will be 8 mm long 1.7 mm diameter titanium screws manufactured by Forestadent and are commercially available and currently widely used in orthodontic treatment in both private practice and educational settings. Since antibiotic prophylaxis is considered the standard of care with traditional dental implants, the investigators believe that such prophylaxis will decrease the failure rate of orthodontic mini-screw implants also.

DETAILED DESCRIPTION:
Subjects will be selected for the study based on treatment plans for Phase II orthodontics at Saint Louis University Center for Advanced Dental Education orthodontics program, which require the use of palatally placed mini-screw implants for anchorage control. If the patient is at or beyond the age of 18 years, they will be approached about this study. If the patient is under the age of 18 years, the parent or legal guardian of the patient will be approached. After the consult is completed, where the treatment plan has been explained and standard consent forms have been signed, a member of the research team will verbally confirm with the patient or the patient and parent/guardian that the patient cannot be excluded from the study based on exclusion criteria from the patient's medical history. Orthodontic treatment at SLU CADE involves monthly visits to the orthodontic clinic where patients receive orthodontic treatment, including leveling and aligning of teeth with archwires and fixed appliances on teeth, space closure, occlusion correction, and finishing and detailing. Mini-screw placement is not necessary nor included in all treatment plans given at SLU CADE orthodontics. The possible subjects for the study will patients who will receive mini-screw implants as a course of their treatment for orthodontic anchorage (standard of care).

Participants will be weighed so that appropriate dosing can be ensured and randomized 1:1 to receive either and antibiotic (Amoxicillin) or a placebo (glucose) 1 hour prior to mini-screw insertion (research related). Patients weighing less than 40 kg will be given 50mg/kg. The Amoxicillin and the placebo (glucose) will be prepared in capsule form by a pharmacist and made to look identical. The Amoxicillin or placebo will be dispensed at CADE and taken at CADE 1 hour prior to the procedure. Standard procedure for dispensing Amoxicillin at SLU CADE is to draw appropriate dosage from the dispensary and provide Amoxicillin to at risk patients prior to invasive dental procedures, in accordance with prophylaxis guidelines set form by the American Heart Association. Documentation of dosage and time of dispensing is noted in the patient record. However, in this study, documentation in the patient dental record will only reflect that either a placebo or Amoxicillin was given as part of a randomized controlled trial. Standard of care for orthodontic mini-screw implants includes oral hygiene instructions and 1 week of oral antibiotic mouth rinse use (.12% Chlorhexidine) and all participants in this study will follow standard of care in addition to the administration of either placebo or antibiotic. Randomization between control or experimental group will be conducted by the Research Chair, Hiroshi Ueno, and the PI will have no knowledge of to which group subjects are assigned.

Participants will be followed at time of mini-screw placement (T0), 1 month post procedure (T1), 3 months post-procedure (T2), and 6 months post-procedure (T3). The participant has standard of care appointments at these time points, so there are not any extra visits for research purposes. At these appointment, participants will undergo an intra-oral exam to determine mobility of the mini-screw(s), to check for inflammation at the site of mini-screw placement, assess oral hygiene at the site of mini-screw placement, and be asked to rate both their pain and tenderness related to the mini-screw. Pain is defined as spontaneous pain frim the mini-screw site. Tenderness is defined as pain resulting from palpation of the mini-screw. Mobility will be determined by placing a small amount of force on the mini-screw with a cotton plier. The amount of mobility will be assessed as having no mobility (Grade 0), having between 0mm and 1 mm of mobility (Grade 1), or having more than 1 mm of mobility (Grade 2). Inflammation will be assessed as having no redness or swelling at the site (Grade 0), having redness only at the site (Grade 1), or having both redness and swelling (Grade 2). Oral hygiene will be assessed as having no visible plaque at the site (Grade 0), having small amounts of plaque at the site (Grade 1), or having moderate to large amounts of plaque at the site (Grade 2). Pain and tenderness will be evaluated separately and will be assessed by asking the patient to rate their pain level on a scale of 0 to 10, 0 being no pain and 10 being unbearable, excruciating pain. A member of the research team will make these evaluations at each time point. All five of these would be assessed as part of the standard of care for mini-screw placement, regardless of participation in the research study or lack thereof. The only action related to the research that is not standard of care is the dispensing of either the antibiotic or the placebo at 1 hour prior to mini-screw placement.

Success of the mini-screw will be defined as number of survival with "Mobility Grade 0 or 1" & "No Pain" & "Inflammation Grade 0 or 1".

Failure of the mini-screw will be immediately determined as failed if the mini-screw is not present at one of the time points or upon an assessment of Grade 2 mobility. Grade 2 mobility will result in removal of the mini-screw.

If the mini-screw implants fail, the participants will have the mini-screw removed. It is up to assigned instructors as to whether or not mini-screws will be replaced. If the mini-screws will not be replaced, the patient will be removed from the study, but all data collected will be included in the research.

Standard of Care will be followed in all instances at time points T(0), T(1), T(2) and T(3).

The dependent variable will be success or failure, while the independent variable will be antibiotic prophylaxis or placebo. Failure will be defined as mobile or lost MSIs, and success will be defined as stability of the MSIs maintained after 6 months. 8mm long, 1.5 mm diameter, palatally placed MSIs provided by a single manufacturer (Forestadent) that are immediately force loaded or delayed in force loading will be included in the study. Data will be analyzed with SPSS for Windows (SPSS Inc., Chicago, Ill). A Chi Square test for independence will be used to determine association, if any, between the two categorical variables. This study will establish an alpha of 0.05 and a beta of 0.08322, and to achieve power of 0.91, a sample size of 100 subjects is the goal for recruiting.

ELIGIBILITY:
Inclusion Criteria: Subjects will be selected for the study based on treatment plans for Phase II orthodontics at SLU CADE orthodontics program, which require the use of palatally placed mini-screw implants for anchorage control.

Exclusion Criteria:

* Patients with experience in previous MSI placements
* allergy to amoxicillin
* allergy to Beta-lactam based antibiotics
* medical syndrome diagnoses
* psychiatric disorders (ADHD, autism, manic-depressive disorder, etc.)
* a compromised immune system
* impaired or decreased kidney function
* Type I or Type II diabetes
* patients taking Probenicid or Allopurinol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Mini-screw implant success or failure | T(0) at time of insertion
  Participants will undergo an intra-oral exam to determine mobility of the mini-screw(s), to check for inflammation at the site of mini-screw placement. Mobility will be determined by placing a small amount of force on the mini-screw with a cotton plier. The amount of mobility will be assessed as having no mobility (Grade 0), having between 0mm and 1 mm of mobility (Grade 1), or having more than 1 mm of mobility (Grade 2). Inflammation will be assessed as having no redness or swelling at the site (Grade 0), having redness only at the site (Grade 1), or having both redness and swelling (Grade 2). Success of the mini-screw will be defined as number of survival with "Mobility Grade 0 or 1" & "No Pain" & "Inflammation Grade 0 or 1".
  Failure of the mini-screw will be immediately determined as failed if the mini-screw is not present at one of the time points or upon an assessment of Grade 2 mobility. Grade 2 mobility will result in removal of the mini-screw.
Mini-screw implant success or failure | T(1) at 1 month post-placement
  Participants will undergo an intra-oral exam to determine mobility of the mini-screw(s), to check for inflammation at the site of mini-screw placement. Mobility will be determined by placing a small amount of force on the mini-screw with a cotton plier. The amount of mobility will be assessed as having no mobility (Grade 0), having between 0mm and 1 mm of mobility (Grade 1), or having more than 1 mm of mobility (Grade 2). Inflammation will be assessed as having no redness or swelling at the site (Grade 0), having redness only at the site (Grade 1), or having both redness and swelling (Grade 2). Success of the mini-screw will be defined as number of survival with "Mobility Grade 0 or 1" & "No Pain" & "Inflammation Grade 0 or 1".
  Failure of the mini-screw will be immediately determined as failed if the mini-screw is not present at one of the time points or upon an assessment of Grade 2 mobility. Grade 2 mobility will result in removal of the mini-screw.
Mini-screw implant success or failure | T(2) at 3 months post-placement
  Participants will undergo an intra-oral exam to determine mobility of the mini-screw(s), to check for inflammation at the site of mini-screw placement. Mobility will be determined by placing a small amount of force on the mini-screw with a cotton plier. The amount of mobility will be assessed as having no mobility (Grade 0), having between 0mm and 1 mm of mobility (Grade 1), or having more than 1 mm of mobility (Grade 2). Inflammation will be assessed as having no redness or swelling at the site (Grade 0), having redness only at the site (Grade 1), or having both redness and swelling (Grade 2). Success of the mini-screw will be defined as number of survival with "Mobility Grade 0 or 1" & "No Pain" & "Inflammation Grade 0 or 1".
  Failure of the mini-screw will be immediately determined as failed if the mini-screw is not present at one of the time points or upon an assessment of Grade 2 mobility. Grade 2 mobility will result in removal of the mini-screw.
Mini-screw implant success or failure | T(3) at 6 months post-placement
  Participants will undergo an intra-oral exam to determine mobility of the mini-screw(s), to check for inflammation at the site of mini-screw placement. Mobility will be determined by placing a small amount of force on the mini-screw with a cotton plier. The amount of mobility will be assessed as having no mobility (Grade 0), having between 0mm and 1 mm of mobility (Grade 1), or having more than 1 mm of mobility (Grade 2). Inflammation will be assessed as having no redness or swelling at the site (Grade 0), having redness only at the site (Grade 1), or having both redness and swelling (Grade 2). Success of the mini-screw will be defined as number of survival with "Mobility Grade 0 or 1" & "No Pain" & "Inflammation Grade 0 or 1".
  Failure of the mini-screw will be immediately determined as failed if the mini-screw is not present at one of the time points or upon an assessment of Grade 2 mobility. Grade 2 mobility will result in removal of the mini-screw.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Ueno, DDS, Study Chair — Full time faculty
Locations (1):
- Saint Louis University Center for Advanced Dental Education, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Background] Berens A, Wiechmann D & Rudiger J. "L'ancrage intra-osseux en orthodontie a' l'aide de mini et de microvis." International Orthodontics (2005) 3: 235-43.
- [Background] Carano A, Melsen B. Implants in orthodontics. Interview. Prog Orthod. 2005;6(1):62-9. No abstract available. English, Italian. PMID 15891785
- [Background] Cope J. "Temporary anchorage devices in orthodontics: a paradigm shift." Seminars in Orthodontics (2005)11:3-9.
- [Background] Costa A, Raffainl M, Melsen B. Miniscrews as orthodontic anchorage: a preliminary report. Int J Adult Orthodon Orthognath Surg. 1998;13(3):201-9. PMID 9835819
- [Background] Esposito M, Grusovin MG, Worthington HV. Interventions for replacing missing teeth: antibiotics at dental implant placement to prevent complications. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD004152. doi: 10.1002/14651858.CD004152.pub4. PMID 23904048
- [Background] Esposito M, Hirsch JM, Lekholm U, Thomsen P. Biological factors contributing to failures of osseointegrated oral implants. (II). Etiopathogenesis. Eur J Oral Sci. 1998 Jun;106(3):721-64. doi: 10.1046/j.0909-8836..t01-6-.x. PMID 9672097
- [Background] Flemmig TF & Newman MG. "Antimicrobials in implant dentistry." In: Newman MG, Kornman K editor. Antibiotics/antimicrobial use in dental practice. Chicago: Quintessence Publishing Co, Inc,(1990):187-200.
- [Background] Freudenthaler JW, Haas R, Bantleon HP. Bicortical titanium screws for critical orthodontic anchorage in the mandible: a preliminary report on clinical applications. Clin Oral Implants Res. 2001 Aug;12(4):358-63. doi: 10.1034/j.1600-0501.2001.012004358.x. English, French, German. PMID 11488865
- [Background] Fritz U, Ehmer A, Diedrich P. Clinical suitability of titanium microscrews for orthodontic anchorage-preliminary experiences. J Orofac Orthop. 2004 Sep;65(5):410-8. doi: 10.1007/s00056-004-0408-x. English, German. PMID 15378195
- [Background] Gray JB, Steen ME, King GJ, Clark AE. Studies on the efficacy of implants as orthodontic anchorage. Am J Orthod. 1983 Apr;83(4):311-7. doi: 10.1016/0002-9416(83)90226-9. PMID 6573144
- [Background] Heymann GC, Tulloch JF. Implantable devices as orthodontic anchorage: a review of current treatment modalities. J Esthet Restor Dent. 2006;18(2):68-79; discussion 80. doi: 10.2310/6130.2006.00013_1.x. PMID 16519871
- [Background] Kanomi R. Mini-implant for orthodontic anchorage. J Clin Orthod. 1997 Nov;31(11):763-7. No abstract available. PMID 9511584
- [Background] Lee SJ, Ahn SJ, Lee JW, Kim SH, Kim TW. Survival analysis of orthodontic mini-implants. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):194-9. doi: 10.1016/j.ajodo.2008.03.031. PMID 20152674
- [Background] Miyawaki S, Koyama I, Inoue M, Mishima K, Sugahara T, Takano-Yamamoto T. Factors associated with the stability of titanium screws placed in the posterior region for orthodontic anchorage. Am J Orthod Dentofacial Orthop. 2003 Oct;124(4):373-8. doi: 10.1016/s0889-5406(03)00565-1. PMID 14560266
- [Background] Odman J, Lekholm U, Jemt T, Branemark PI, Thilander B. Osseointegrated titanium implants--a new approach in orthodontic treatment. Eur J Orthod. 1988 May;10(2):98-105. doi: 10.1093/ejo/10.2.98. No abstract available. PMID 3164683
- [Background] Ohmae M, Saito S, Morohashi T, Seki K, Qu H, Kanomi R, Yamasaki KI, Okano T, Yamada S, Shibasaki Y. A clinical and histological evaluation of titanium mini-implants as anchors for orthodontic intrusion in the beagle dog. Am J Orthod Dentofacial Orthop. 2001 May;119(5):489-97. doi: 10.1067/mod.2001.114300. PMID 11343020
- [Background] Papadopoulos MA, Tarawneh F. The use of miniscrew implants for temporary skeletal anchorage in orthodontics: a comprehensive review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 May;103(5):e6-15. doi: 10.1016/j.tripleo.2006.11.022. Epub 2007 Feb 21. PMID 17317235
- [Background] Prophylaxis in surgery. Veterans Administration Ad Hoc Interdisciplinary Advisory Committee on Antimicrobial Drug Usage. JAMA. 1977 Mar 7;237(10):1003-8. No abstract available. PMID 319261
- [Background] Reynders R, Ronchi L, Bipat S. Mini-implants in orthodontics: a systematic review of the literature. Am J Orthod Dentofacial Orthop. 2009 May;135(5):564.e1-19; discussion 564-5. doi: 10.1016/j.ajodo.2008.09.026. PMID 19409331
- [Background] Roberts WE, Helm FR, Marshall KJ, Gongloff RK. Rigid endosseous implants for orthodontic and orthopedic anchorage. Angle Orthod. 1989 Winter;59(4):247-56. doi: 10.1043/0003-3219(1989)0592.0.CO;2. PMID 2688486
- [Background] Roberts WE, Marshall KJ, Mozsary PG. Rigid endosseous implant utilized as anchorage to protract molars and close an atrophic extraction site. Angle Orthod. 1990 Summer;60(2):135-52. doi: 10.1043/0003-3219(1990)0602.0.CO;2. PMID 2344070
- [Background] Roberts WE, Smith RK, Zilberman Y, Mozsary PG, Smith RS. Osseous adaptation to continuous loading of rigid endosseous implants. Am J Orthod. 1984 Aug;86(2):95-111. doi: 10.1016/0002-9416(84)90301-4. PMID 6589962
- [Background] Sharaf B, Jandali-Rifai M, Susarla SM, Dodson TB. Do perioperative antibiotics decrease implant failure? J Oral Maxillofac Surg. 2011 Sep;69(9):2345-50. doi: 10.1016/j.joms.2011.02.095. Epub 2011 Jun 15. PMID 21676512
- [Background] Wehrbein H, Merz BR. Aspects of the use of endosseous palatal implants in orthodontic therapy. J Esthet Dent. 1998;10(6):315-24. doi: 10.1111/j.1708-8240.1998.tb00510.x. PMID 10321202